CLINICAL TRIAL: NCT05056896
Title: ASPIRED-XT: ASPirin Intervention for the REDuction of Colorectal Cancer Risk -EXTension
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Andrew T. Chan, MD, MPH, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 21-376; R01CA243454 (NIH); R01CA257523 (NIH); R35CA253185-01 (NIH); K01DK120742-01A1 (NIH)
Record Dates: First submitted 2021-09-15; First posted 2021-09-27 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Colorectal Cancer
Keywords: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-Blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Low Dose Aspirin (Experimental): Participants will be randomly assigned to aspirin group and receive a daily low dose aspirin (81 mg) for the duration of the study up to 12 weeks.
  Interventions: Drug: Aspirin
- Placebo (Experimental): Participants will be randomly assigned to placebo group and receive a daily placebo capsule for the duration of the study up to 12 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Aspirin — Capsule taken orally
  Other Names: acetylsalicylic acid (ASA); Salicylic Acid Acetate
  Arms: Low Dose Aspirin
Other: Placebo — Capsule taken orally
  Arms: Placebo

SUMMARY:
This research study is studying a drug intervention as a possible chemoprevention strategy for colorectal cancer.

The name of the study intervention involved in this study is:

* Low Dose Aspirin

DETAILED DESCRIPTION:
This is prospective, double-blind, placebo-controlled, randomized clinical trial to measure the effects of daily low-dose (81 mg/day) aspirin on tissue, urine, plasma, and stool biomarkers associated with colorectal cancer with a focus on the effect of age. It is a direct extension of an earlier study: ASPIRED trial NCT02394769

Aspirin is part of the non-steroidal anti-inflammatory drug (NSAID) family, which are drugs routinely used for their pain-killing (analgesic), fever-reducing (antipyretic), or anti-inflammatory properties. Most NSAIDs are available as over-the-counter formulations. Substantial evidence has conclusively demonstrated that aspirin reduces the risk of colorectal polyps and cancer, yet there remains uncertainty surrounding its mode of action. Aspirin may prevent colorectal cancer through multiple interrelated biological mechanisms including the reduction of chronic inflammation, a known risk factor for colorectal cancer. Aspirin has been shown to directly affect prostaglandins, a class of biologic molecules that play important roles in controlling the normal inflammatory responses within your body. The exact mechanism by which aspirin acts to prevent colorectal cancer is still unknown.This study is looking at the mechanisms of aspirin's anti-cancer effect, which may lead to the discovery of novel specific characteristics (markers) that can be used to select patients for aspirin treatment. the study will also look at the effect age may have on these mechanisms.

The research study procedures include screening for eligibility and study treatment and scheduling two clinical research visits immediately before and after intervention with the study drug.

Participants will be randomized into two groups.

* Arm A: Daily Placebo (no aspirin) for the duration of the study.
* Arm B: Daily low dose aspirin (81 mg/day) for the duration of the study.

Participants may be contacted periodically after the study (no more than 1- 2 times annually) for up to 10 years to follow-up on additional information including any continued aspirin use or follow-up colonoscopy results.

It is expected that about 160 people will take part in this research study.

The National Cancer Institute (NCI) of the National Institutes of Health (NIH) is supporting this research study by providing funding for the research study.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have undergone screening or surveillance colonoscopy with removal of at least one adenoma within the last 9 months.
* Age greater than or equal to 18 years and less than 55 years or greater than or equal to 65 years at the time of enrollment This study will only include adult participants because colorectal carcinogenesis in children is more likely to be related to a cancer predisposition syndrome with distinct biological mechanisms compared with sporadic colorectal cancer in adults.
* ECOG performance status ≤2 (Karnofsky ≥60%, see Appendix A).
* Not currently taking aspirin (any dose) within the last 6 months.
* The effects of aspirin on the developing human fetus are unknown. For this reason, women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she is participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Use of any non-aspirin non-steroidal anti-inflammatory drug (NSAID) at any dose at least three times a week during the two months prior to randomization.
* Diagnosis of inflammatory bowel disease, liver or kidney disease, bleeding diathesis.
* Any prior diagnosis of gastrointestinal cancer (including esophageal, small intestine, colon, pancreatic), or any diagnosis of other cancers (with the exception of non-melanoma skin) in which there has been any active treatment within the last three years.
* Participants who are receiving any other investigational agents.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to aspirin.
* Known diagnosis of Familial Adenomatous Polyposis (FAP) or Hereditary Non-Polyposis Colorectal Cancer (HNPCC, Lynch Syndrome).
* Any adenoma that was not completely removed during previous colonoscopy.
* History of aspirin intolerance, bleeding diathesis, peptic ulcer or gastrointestinal bleed, endoscopic complications, or contraindication to colonoscopy.
* Inability or unwillingness to abstain from non-protocol use of aspirin or NSAIDs or to provide blood, urine, or stool samples or colon biopsies during the study.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant or breastfeeding. Pregnant women are excluded from this study because aspirin is an FDA Category D agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with aspirin, breastfeeding should be discontinued if the mother is treated with aspirin.
* Participant must be able to swallow pills.
* Participant is taking any anticoagulant agent (e.g. warfarin) or antiplatelet agent (e.g. clopidogrel).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2022-06-03 (Actual); Primary Completion 2024-11-27 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of ISC marker gene expression | 2 months
  Assess the difference in the change of ISC marker using scRNA-seq data analysis

SECONDARY OUTCOMES:
Change in Urinary PGE-M | 2 months
  Comparing change in PGE-M between treatment groups (aspirin and placebo) using a two-sample t-test.
Change in urinary Plasma GDF-15 | 2 months
  Comparing change inGDF-15 between aspirin and placebo groups, using a two-sample t-test.
ChIP-seq Analysis of Colonic Epithelium | 2 months
  Analysis of the ChIP-seq data (>60 million reads, 50-bp paired end) using the publicly available Cistrome Analysis Pipeline
Gene Expression Analysis of Colonic Epithelium | 2 months
  RNA-seq sequence data (> 50 million reads) will be mapped to hg19 through use of TopHat2.
Change in Microbiome | 2 months
  Aspirin use and dose will be associated with microbial operational taxonomic units (OTUs) using the Biobakery3 computational analysis pipeline.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew T Chan, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital Cancer Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation